CLINICAL TRIAL: NCT07337447
Title: PRODIGE 113 (FFCD 2314) - REWENEC 01 STUDY Randomized Trial of FOLFIRI + Zimberelimab + Domvanalimab vs FOLFIRI With a Hybrid Synthetic Control Arm in Second Line Treatment of Neuroendocrine Carcinoma of Gastro-enteropancreatic or Unknown Origin. Phase II Comparative Randomized Study - Multicentric
Brief Title: Trial of FOLFIRI + Zimberelimab + Domvanalimab vs FOLFIRI With a Hybrid Synthetic Control Arm in Second Line Treatment of Neuroendocrine Carcinoma of Gastro-enteropancreatic or Unknown Origin (REWENEC 01)
Acronym: REWENEC 01
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Collaborators: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 69HCL24_0759; 2024-519922-19-00 (EU CTIS Number)
Record Dates: First submitted 2025-12-08; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Carcinoma, Neuroendocrine
Keywords: Carcinoma, Neuroendocrine; gastro-enteropancreatic or unknown origin; GEP/UK NEC
MeSH Terms: conditions — Carcinoma, Neuroendocrine | interventions — zimberelimab; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental arm (EA) 61 patients prospectively enrolled to receive the experimental treatment in th (Experimental): FOLFIRI every 14 days + Zimberelimab IV every 28 days + Domvanalimab UV every 28 days
  Interventions: Drug: FOLFIRI + Zimberelimab + Domvanalimab
- Hybrid Synthetic Control Arm (HSCA) combines historical data from 45 patients in the BEVANEC trial a (Active Comparator): 45 patients in this group from the BEVANEC trial and 16 patients in this group will be prospectively enrolled and will receive FOLFIRI every 14 days IV every 28 days
  Interventions: Drug: FOLFIRI (standard of care)

INTERVENTIONS:
Drug: FOLFIRI + Zimberelimab + Domvanalimab — FOLFIRI every 14 days + Zimberelimab IV every 28 days + Domvanalimab IV every 28 days
  Arms: Experimental arm (EA) 61 patients prospectively enrolled to receive the experimental treatment in th
Drug: FOLFIRI (standard of care) — FOLFIRI every 14 days IV every 28 days
  Arms: Hybrid Synthetic Control Arm (HSCA) combines historical data from 45 patients in the BEVANEC trial a

SUMMARY:
Background Neuroendocrine carcinomas (NECs) of gastro-entero-pancreatic (GEP) or unknown (UK) origin are rare and highly aggressive diseases. The recommended first-line (L1) treatment is platinum-etoposide combination therapy, which has a progression-free survival (PFS) of only 4-9 months and a median overall survival (OS) of approximately 12 months. All patients experience relapse, often rapidly after this first line of chemotherapy. The standard second-line (L2) chemotherapies recommended by ESMO, ENETS, and NCCN, FOLFIRI and FOLFOX, have modest efficacy with a PFS of 3 months and a median OS of 6 months. The BEVANEC study (PHRCK 2014, NCT02820857) reported no benefit of FOLFIRI + bevacizumab compared to FOLFIRI in a randomized phase II study that enrolled 150 patients in 26 centers over a period of 5 years in France.

To date, the most promising efficacy data for this highly aggressive cancer come from clinical trials of immune checkpoint inhibitors (ICIs) targeting the PD-1/PD-L1 checkpoint. For example, in France, the non-comparative phase II NIPINEC trial (NCT03591731) randomized patients to receive nivolumab +/- ipilimumab in L2/3 and achieved its primary evaluation criterion (ORR-8 weeks>10%). Other trials in Europe and worldwide have also reported efficacy data in the context of single-arm studies.

Scientific Questions and Unmet Needs:

1. New therapeutic options/perspectives are necessary for patients with GEP/UK NECs given the limited overall survival.
2. Approximately 50% of patients experienced early progression under immunotherapy in the NIPINEC trial and other trials, which may be explained by the absence of chemotherapy combined with immunotherapy and/or the existence of resistance mechanisms.
3. In the GEP/UK NEC indication, the design of these immunotherapy trials has been non-comparative single-arm studies because the realization of randomized comparative trials is considered very difficult for these very rare cancers (incidence <5/million).

Rationale for the REWENEC-01 Trial The DURIGAST PRODIGE 59 study, conducted by the FFCD, demonstrated the feasibility and safety of the FOLFIRI + double immune checkpoint inhibitor (anti-PD-1 and anti-CTLA4) combination, as well as for the combination Folfox-Domvanalimab-Zimberelimab (anti-PD-1 and anti-TIGIT). In a translational study of the immune phenotype in patients with NECs treated with the anti-PD1 pembrolizumab, an increase in TIGIT expression was observed after pembrolizumab treatment and higher TIGIT expression on T cells in the blood of patients with high Ki67 expression in their tumors. These data suggest that TIGIT is a potential complementary therapeutic target to PD-1/PD-L1 checkpoint inhibition in GEP/UK NECs. Domvanalimab has been developed as an anti-TIGIT monoclonal antibody and zimberelimab as an anti-PD-1.

Design and primary objective of the REWNEC-01 Trial The REWENEC-01 trial is a comparative phase II trial that will randomize GEP/UK NEC patients between an experimental arm FOLFIRI+Zimberelimab + Domvanalimab and a control arm FOLFIRI in L2. The FOLFIRI arm will be a "hybrid" synthetic control arm composed of patients from historical/external data from the FOLFIRI arm of BEVANEC and French retrospective studies RBNEC and CEPD, mixed with patients recruited prospectively during the trial and randomized to the control arm. The randomization ratio for patients included prospectively during the trial will be 4:1 (4 patients assigned to FOLFIRI+Zimberelimab + Domvanalimab for 1 patient assigned to FOLFIRI). The randomization algorithm will take into account "external" patients assigned progressively to the control arm to obtain a 1:1 ratio between the trial arms, with balanced distributions of stratification factors between the two arms.

With 77 patients to be included, this strategy will provide statistical power equivalent to that of a trial including 122 patients, sufficient to demonstrate an advantage in overall survival rate at 12 months from 32% to 50%.

The hypotheses related to efficacy criteria are formulated a priori, as recommended by the FDA guidance document on trials with synthetic/external control arms. The proof of concept has been reported at ESMO 2023. The primary judgment criterion will be the overall survival rate at 12 months because it is a strong and significant criterion for translating the clinical benefit of the Chemotherapy + Zimberelimab + Domvanalimab combination. The design with a hybrid synthetic control arm allows for the consideration of a randomized comparative study in a cancer as rare as neuroendocrine carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged ≥ 18 years old,
* Poorly differentiated neuroendocrine carcinoma (NEC) [or mixed tumor with NEC component is > 30%, the patient is eligible] with ki 67 > 20% from a gastrointestinal tract (from esophagus to anal canal) or biliopancreatic primary or an unknown primary cancer, locally advanced and/or metastatic,
* Centralized review of the diagnostic by a consulting pathologist specialized in NET (TENPATH network),
* Recommendation of a second-line chemotherapy after progression (documented using the RECIST criteria v.1.1) and after a first-line chemotherapy treatment by cisplatin (or carboplatin) + etoposide or in the event of progression in the 6 months following the discontinuation of this first-line treatment,
* Patient presenting at least one measurable target lesion according to the RECIST criteria v.1.1, in an area not previously irradiated,
* General condition ≤ 1 (ECOG-PS),
* Patient of childbearing age accepting to use a highly effective method of contraception during treatment and until 6 months after discontinuation of chemotherapy and 4 months after the last dose of domvanalimab and zimberelimab. Men sexually active must agree to use a highly effective method of contraception during treatment and for at least 6 months after discontinuation of chemotherapy and 4 months after the last dose of domvanalimab and zimberelimab,
* Patient who signed the informed consent form.
* Patient affiliated to National French social security system

Exclusion Criteria:

* Well differentiated neuroendocrine tumor whatever the grade,
* First-line chemotherapy other than cisplatin (or carboplatin) and etoposide,
* Prior immunotherapy,
* Prior malignancy active within the previous 2 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix, breast, or prostate cancer,
* Pregnant or breastfeeding woman,
* Lack of efficient contraception (for men or women of reproductive age),
* All medical, geographical, social, and psychological conditions or a legal situation that will not allow the patient to finish the study or sign an informed consent form,
* Patient with asymptomatic brain metastasis or with previously treated brain metastasis relating to the study drugs
* Any of the following uncontrolled progressive diseases in the 6 months before randomization: liver failure, renal insufficiency, respiratory distress, congestive heart failure (NYHA III-IV), unstable angina, myocardial infarction, significant arrhythmia,
* Partial and complete dihydropyrimidine dehydrogenase (DPD) deficiency: uracil level ≥ 16 ng/ml,
* Known Gilbert's syndrome,
* Total bilirubin level >1.5 x the upper limit of normal (ULN); ASAT and/or ALAT > 5 x ULN; TP < 50 % (Except for patient's treated with Vitamin K antagonists or direct oral anticoagulants with INR <3 ),
* Neutrophils <1.5x109/l, platelets <100x109/l, hemoglobin < 9 g/dl,
* Chronic uncontrolled diarrhea, unresolved intestinal occlusion or subocclusion,
* History of anaphylactic reaction or known intolerance to atropine (sulfate) or to loperamide or to antiemetics administered in association with Folfiri,
* All treatment with concomitant anticonvulsive agents, CYP3A4 inducers (phenytoin, phenobarbital, carbamazepine); patients with these treatments should have stopped them, for at least 7 days before inclusion in the study,
* Chronic medical condition requiring the ongoing use of supra-physiologic doses of systemic corticosteroids (>10 mg/day of oral prednisone or equivalent) or systemic immunosuppressive medications. Immunosuppressive medications, including chronic systemic corticosteroids at supraphysiologic doses should have been stopped 14 days before the first dose (except for participants who require hormone replacement therapy such as hydrocortisone).
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* History of (non-infectious) pneumonitis that required steroids, or current pneumonitis.
* History of severe hypersensitivity reaction to any monoclonal antibody (mAb) therapy.
* Live attenuated vaccines within 28 days prior enrolment.
* Any concurrent anticancer therapy, including chemotherapy, radiotherapy (except palliative radiotherapy), immunotherapy, biologic, or hormonal treatment. Concurrent use of hormones for noncancer-related conditions is permitted.
* Known hypersensitivity to any investigational product (IP), or any excipient contained in the formulations of the study interventions.
* Known immunodeficiency or human immunodeficiency virus (HIV) infection with HIV viral load ≥200 copies/mL or CD4+ T-cell count <350 cells/μL, or taking medications that may interfere with metabolism of study drugs.
* Known acute hepatitis B, known chronic hepatitis B infection with active untreated disease, or known active hepatitis C infection. In participants with a history of HBV or HCV, participants with detectable viral loads will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival (%) between FOLFIRI and FOLFIRI+Zimberelimab+Domvanalimab | 6 months after the start of treatment 12 months after the start of treatment
  Length of time from randomization that patients included in the study are still alive. Analyzed in modified intention to treat

SECONDARY OUTCOMES:
Progression free survival (PFS) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from randomization to disease progression or death, whatever the cause. Alive and no progressive patients at last follow-up will be considered as censored
Overall response rate (ORR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  local radiological evaluation using RECIST 1.1
Duration of response (DoR) | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Time from response (complete or partial) to progression or death, estimated in patients who reached a response and are RECIST 1.1 evaluable
Disease control rate | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Defined as the proportion of RECIST 1.1 evaluable patients in objective response or with stable disease.
Evaluation of toxicity | At the Day 1 of each cycles (each cycle is 4 weeks)
  assessed by NCI CTCAsE v5.0
Evaluation of toxicity | at the Day 15 of each cycles (each cycle is 4 weeks)
  assessed by NCI CTCAsE v5.0
Questionnaire Quality of life QLQ-C30 | at the day 1 of Cycle 2 (1 cycle is 4 weeks)
  Questionnaire QLQ-C30
Questionnaire Quality of life EQ 5D-5L | at the day 1 of Cycle 2 (1 cycle is 4 weeks)
  Questionnaire EQ 5D-5L
Questionnaire Quality of life | Every 8 weeks through study completion, an average of 2 years
  Questionnaire QLQ-C30
Questionnaire Quality of life | Every 8 weeks through study completion, an average of 2 years
  Questionnaire EQ 5D-5L

CONTACTS AND LOCATIONS:
Overall Officials: Thomas WALTER, MD, Principal Investigator — Hospices Civils de Lyon
Locations (21):
- France (21):
  - CHU Amiens Picardie, Amiens
  - CHU Avicenne APHP, Bobigny
  - CHU Caen Normandie, Caen
  - Hôpital Beaujon, Clichy
  - Hôpital Henri MONDOR, Créteil
  - CHU Dijon, Dijon
  - CHU de Grenoble, Grenoble
  - Centre Oscar Lambret, Lille
  - Service d'Oncologie Médicale - Hôpital Edouard Herriot - Hospices Civils de Lyon, Lyon
  - CHU Timone, Marseille
  - Institut Paoli Calmettes, Marseille
  - CHU Montpellier - Hôpital Saint Eloi, Montpellier
  - HEGP, Paris
  - Hôpital Saint Antoine APHP, Paris
  - Hôpital Saint Louis APHP, Paris
  - CHU de Bordeaux - Hôpital Haut-Leveque, Pessac
  - CHU de Poitiers, Poitiers
  - Hôpital Robert Debré, CHU de Reims, Reims
  - CHU Rouen, Rouen
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif